CLINICAL TRIAL: NCT07222748
Title: A Phase 3, Randomized, Double-blind, Comparator- and Placebo-controlled Study to Evaluate the Safety and Efficacy of TLC590 for Postsurgical Pain Management Following Bunionectomy
Brief Title: A Study of TLC590 for Postsurgical Pain Following Bunionectomy
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: TLC Biopharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Taiwan Liposome Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TLC590A3004
Record Dates: First submitted 2025-10-28; First posted 2025-10-30 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Postoperative Pain
Keywords: Bunion; Bunionectomy; Bunion surgery; Postoperative pain
MeSH Terms: conditions — Pain, Postoperative; Bunion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- TLC590 (Experimental)
  Interventions: Drug: TLC590
- Liposomal Bupivacaine (Active Comparator)
  Interventions: Drug: Liposomal Bupivacaine
- Saline Placebo (Placebo Comparator)
  Interventions: Drug: Saline Placebo

INTERVENTIONS:
Drug: TLC590 — TLC590 (Ropivacaine Extended-Release Injectable Suspension)
  Arms: TLC590
Drug: Liposomal Bupivacaine — Bupivacaine Liposome Injectable Suspension
  Arms: Liposomal Bupivacaine
Drug: Saline Placebo — Normal Saline 0.9%
  Arms: Saline Placebo

SUMMARY:
This is a Phase 3, randomized, double-blind, comparator- and placebo-controlled study to evaluate analgesic efficacy and safety of TLC590 via local infiltration in adult subjects following bunionectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide written informed consent.
2. Male or female aged 18 years or older (inclusive).
3. Scheduled to undergo a primary unilateral, transpositional first metatarsal bunionectomy with osteotomy and internal fixation under regional anesthesia.
4. ASA Physical Status Classification of 1 or 2.
5. Male subjects must be either biologically or surgically sterile or commit to the use of a reliable method of birth control (must agree to use double-barrier contraception in the event of sexual activity) or be practicing abstinence.
6. Female subjects are eligible only if not pregnant, not lactating, not planning to become pregnant during the study, or committing to the use of a highly effective method of birth control.
7. BMI >18 ~ ≤39 kg/m2, with a minimum weight of 50 kg.

Exclusion Criteria:

1. An abnormal clinical laboratory test value.
2. Evidence of a clinically significant abnormal 12-lead ECG.
3. History of orthostatic hypotension, syncope, or other syncopal attacks.
4. History or any clinical manifestation of significant renal, hepatic, gastrointestinal, cardiovascular, metabolic, neurologic, psychiatric, or other conditions that have been assessed by the Investigator to make the subject unsuitable for participation in the study.
5. History of seizures or taking anticonvulsants.
6. History of cardiac arrhythmia or taking Class III antiarrhythmic drugs.
7. History of sleep apnea or at-home CPAP treatment.
8. History of hypersensitivity to ropivacaine, bupivacaine, any other amide-type local anesthetic, or any other trial-required medications.
9. History of severe or refractory PONV due to other etiologies, including, but not limited to gastric outlet obstruction, hypercalcemia, or active peptic ulcer, deemed clinically significant by the Investigator.
10. Any lifetime history of a suicidal attempt or any suicidal behavior.
11. History or positive test results of HIV, HCV, or HBV.
12. History or current report of substance abuse including illicit drug abuse and/or alcohol abuse.
13. Positive results on the urine drug screen or alcohol breath test.
14. Pre-existing concurrent acute, or chronic painful restrictive/physical condition that may confound postoperative pain assessments or is expected to require analgesic treatment during the study.
15. Has known or suspected daily use of opioids for longer than 4 days per week within 6 months.
16. Use of daily analgesics for longer than 4 days per week for a chronically painful condition.
17. Is receiving oxygen therapy.
18. Use of any of the pre-specified medications prior to the study surgical procedure or as specified.
19. Malignancy in the past 2 years, except for non-metastatic basal cell or squamous cell carcinoma of the skin or localized carcinoma in situ of the cervix.
20. Personal or family history of malignant hyperthermia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-11-17 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Mean Area Under the Curve (AUC) of the Numeric Rating Scale (NRS) Pain Intensity Scores Through 72 Hours Postsurgery (AUC0-72), Compared with Saline Placebo. | 72 hours
  Pain intensity is measured using an 11-point Numeric Rating Scale (NRS) (0-10), where 0 represents "no pain" and 10 represents "worst pain imaginable", and higher scores indicate worse pain.

SECONDARY OUTCOMES:
Proportion of subjects who are opioid-free for TLC590 compared with Saline Placebo. | 72 hours
Mean Area Under the Curve (AUC) of the Numeric Rating Scale (NRS) Pain Intensity Scores Through 72 Hours Postsurgery (AUC0-72), Compared with Bupivacaine Liposome. | 72 hours
  Pain intensity is measured using an 11-point Numeric Rating Scale (NRS) (0-10), where 0 represents "no pain" and 10 represents "worst pain imaginable", and higher scores indicate worse pain.
Mean Total Postoperative Opioid Consumption for TLC590 Compared with Saline Placebo | 72 hours
Proportion of subjects who are opioid-free for TLC590 compared with Bupivacaine Liposome. | 72 hours
Mean Total Postoperative Opioid Consumption for TLC590 Compared with Bupivacaine Liposome. | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Tien-Tzu Tai, MD, Study Director — Taiwan Liposome Company
Locations (4):
- United States (4):
  - Clinical Pharmacology of Miami, Miami, Florida
  - First Surgical Hospital, Bellaire, Texas
  - Memorial Hermann Village, Houston, Texas
  - Endeavor Clinical Trials, San Antonio, Texas